CLINICAL TRIAL: NCT03770000
Title: An Open Label, Phase I/II Study to Evaluate the Safety and Efficacy of Tenalisib (RP6530), a Novel PI3K δ/γ Dual Inhibitor Given in Combination With a Histone Deacetylase (HDAC) Inhibitor, Romidepsin in Adult Patients With Relapsed/Refractory T-cell Lymphoma
Brief Title: Safety and Efficacy of Tenalisib (RP6530) in Combination With Romidepsin in Patients With Relapsed/Refractory T-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP6530+Romidepsin-1805
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: T Cell Lymphoma
Keywords: T cell Lymphoma; RP6530; Tenalisib; Romidepsin
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — tenalisib; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tenalisib+Romidepsin (Experimental): Participants receive Tenalisib in escalating doses daily Orally BID and Romidepsin in escalating doses intravenously on day 1, 8 and 15
  Interventions: Drug: Tenalisib; Drug: Romidepsin

INTERVENTIONS:
Drug: Tenalisib — Tenalisib, BID orally daily
  Other Names: RP6530
Drug: Romidepsin — Romidepsin IV

SUMMARY:
To characterize safety, tolerability and to establish the maximum tolerated dose (MTD) of Tenalisib in combination with Romidepsin in patients with R/R T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed T-cell lymphomas at the enrolling institution.
2. Disease status as defined as relapsed or progressed patients who have received at least one systemic therapy.
3. The patients should have received NOT more than three prior systemic combination chemotherapies
4. PTCL patients must have measurable disease defined as at least one bidimensional measurable lesion with minimum measurement of > 1.5 cm in the longest diameter.
5. Must have ECOG performance status ≤ 2
6. Adequate bone marrow, liver and renal function in line with below mentioned laboratory requirements.

   1. Hemoglobin ≥8.0 g/dL
   2. Absolute neutrophil count (ANC) ≥1,000/µL
   3. Platelet count ≥75,000/μL
   4. Total bilirubin ≤1.5 times the ULN (or ≤3 x ULN, if patient has Gilbert syndrome)
   5. AST (SGOT) and ALT (SGPT) ≤ 3 x ULN; ≤ 5 ULN in case of liver involvement
   6. Calculated creatinine clearance (CrCl) > 50 ml/min by Cockcroft-Gault formula
7. Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential.
8. Provide written informed consent prior to any study-specific screening procedures.
9. Willingness and capability to comply with the requirements of the study

Exclusion Criteria:

1. Patient receiving anticancer therapy including any investigational therapy ≤3 weeks or 5 half-lives (whichever is shorter) prior to C1D1.
2. Patient who discontinued prior therapy with PI3K inhibitors or HDAC inhibitors due to drug toxicity.
3. PTCL patients with Allo-SCT on active GVHD or immunosuppression therapy within 3 months prior to C1D1. CTCL patients with the history of Allo-SCT will be excluded.
4. Patient with medical conditions requiring the use of systemic immunosuppressive medications (> 20 mg/day of prednisone or equivalent).
5. Severe bacterial, viral or mycotic infection requiring systemic treatment.
6. Known seropositive requiring anti-viral therapy for human immunodeficiency virus (HIV) infection.
7. Known seropositive requiring anti-viral therapy for hepatitis B virus (HBV) infection OR evidence of active hepatitis B infection as defined by detectable viral load if the antibody tests are positive..
8. Known seropositive requiring anti-viral therapy for hepatitis c virus (HCV) infection OR patients with positive hepatitis C virus Ab.
9. Subjects with active EBV unrelated to underlying lymphoma (positive serology for anti- EBV VCA IgM antibody and negative for anti-EBV EBNA IgG antibody, or clinical manifestations and positive EBV PCR consistent with active EBV infection.
10. Subject with active CMV (positive serology for anti-CMV IgM antibody and negative for anti-CMV IgG antibody and positive CMV PCR with clinical manifestations consistent with active CMV infection) and requiring therapy.
11. Uncontrolled or significant cardiovascular disease including, but not limited to:

    * Congenital long QT syndrome.
    * QTcF interval > 450 msec
    * Myocardial infarction or stroke/TIA within the past 6 months
    * Uncontrolled angina within the past 3 months
    * Significant ECG abnormalities including 2nd degree atrio- ventricular (AV) block (AV) block type II, 3rd degree AV block.
    * History of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation or torsades de pointes),
    * History of other clinically significant heart disease (ie, cardiomyopathy, congestive heart failure with NYHA functional classification III-IV, pericarditis, significant pericardial effusion)
    * Requirement for daily supplemental oxygen therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Hellen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami-Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Rush University Cancer Center, Chicago, Illinois
  - The University of Kansas Cancer Center, Fairway, Kansas
  - Norton Cancer Institute, St Matthews Campus, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center,, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iyer SP, Huen A, Ai WZ, Jagadeesh D, Lechowicz MJ, Okada C, Feldman TA, Ghione P, Alderuccio JP, Champion R, Kim SH, Mohrbacher A, Routhu KV, Barde P, Nair AM, Haverkos BM. Safety and efficacy of tenalisib in combination with romidepsin in patients with relapsed/refractory T-cell lymphoma: results from a phase I/II open-label multicenter study. Haematologica. 2024 Jan 1;109(1):209-219. doi: 10.3324/haematol.2022.281875. PMID 37439343

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose escalation_Cohort 1: RP6530 was administered at 400 mg BID orally daily and Romidepsin was administered at 12 mg/m2, IV on day 1, 8 and 15
- Dose escalation_Cohort 2: RP6530 was administered at 600 mg BID orally daily and Romidepsin was administered at 12 mg/m2, IV on day 1, 8 and 15
- Dose escalation_Cohort 3; Dose expansion_Group 2 (CTCL): RP6530 was administered at 800 mg BID orally daily and Romidepsin was administered at 14 mg/m2, IV on day 1, 8 and 15
- Dose expansion_Group 1 (PTCL): RP6530 was administered at 800 mg BID orally daily and Romidepsin was administered at 12 mg/m2, IV on day 1, 8 and 15
Period: Overall Study
Arm/Group | Dose escalation_Cohort 1 | Dose escalation_Cohort 2 | Dose escalation_Cohort 3 | Dose expansion_Group 1 (PTCL) | Dose expansion_Group 2 (CTCL)
Started | 3 | 3 | 3 | 12 | 12
Completed | 3 | 3 | 2 | 9 | 10
Not Completed | 0 | 0 | 1 | 3 | 2
Not completed — Premature discontinuation due to PD | 0 | 0 | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Dose expansion_Group 1 (PTCL); Dose expansion_Group 2 (CTCL): RP6530 was administered at 800 mg BID orally daily and Romidepsin was administered at 14 mg/m2, IV on day 1, 8 and 15
- Total: Total of all reporting groups
Arm/Group | Dose escalation_Cohort 1 | Dose escalation_Cohort 2 | Dose escalation_Cohort 3 | Dose expansion_Group 1 (PTCL) | Dose expansion_Group 2 (CTCL) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 12 | 12 | 33
Age, Continuous [Median (Full Range); unit: years] | 69.79 [56.53 to 79.44] | 55.72 [49.17 to 66.21] | 49.03 [48.76 to 63.27] | 67.62 [42.89 to 83.44] | 69.67 [61.54 to 80.55] | 66.21 [42.89 to 83.44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 6 | 7 | 16
  Male | 3 | 2 | 1 | 6 | 5 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2 | 4
  White | 2 | 3 | 1 | 11 | 10 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 12 | 12 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Without Dose Limiting Toxicities (DLTs)
Description: The DLTs will be classified according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Time Frame: 28 days
Population: DLT assessment performed in patients who participated in dose escalation phase; A toxicity will be considered dose-limiting if it occurs during the first cycle (4-weeks) of treatment with Tenalisib and Romidepsin combination and is considered related to combination.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose escalation_Cohort 1 | Dose escalation_Cohort 2 | Dose escalation_Cohort 3 | Dose expansion_Group 1 (PTCL) | Dose expansion_Group 2 (CTCL)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
Participants
  No.of Participants with Dose Limiting Toxicities | 0 | 0 | 0 | 0 | 0
  No.of Participants without Dose Limiting Toxicities | 3 | 3 | 3 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR) With Tenalisib and Romidepsin Combination
Description: Overall response (ORR) = CR + PR) was assessed according to the Lugano classification with PTCL and according to the modified Severity Weighted Assessment Tool (mSWAT)/Global assessment in patients with CTCL.
Time Frame: 12 weeks
Population: Patients were considered for efficacy analysis as per protocol only if they had one post treatment efficacy assessment at C3D1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose escalation_Cohort 1 | Dose escalation_Cohort 2 | Dose escalation_Cohort 3 | Dose expansion_Group 1 (PTCL) | Dose expansion_Group 2 (CTCL)
Number analyzed (Participants) | 3 | 3 | 2 | 9 | 10
Participants | 2 | 2 | 0 | 7 | 6

3. Secondary Outcome: Duration of Response (DoR) With Tenalisib and Romidepsin Combination
Description: The time period from the response achieved in patient until the disease progression
Time Frame: 28 weeks
Population: Duration of Response (DoR) is defined as the time when the measurement criteria are first met for PR or CR (whichever is reported first) until the date of documented disease progression or death. Overall number of Participants analyzed for DoR will be the participants who met response as CR or PR
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Dose escalation_Cohort 2: RP6530 was administered at 600 mg BID orally daily and Romidepsin was administered at 14 mg/m2, IV on day 1, 8 and 15
- Dose expansion_Group1 (PTCL Patients); Dose expansion_Group2 (CTCL Patients): RP6530 was administered at 800 mg BID orally daily and Romidepsin was administered at 14 mg/m2, IV on day 1, 8 and 15
Arm/Group | Dose escalation_Cohort 1 | Dose escalation_Cohort 2 | Dose escalation_Cohort 3 | Dose expansion_Group1 (PTCL Patients) | Dose expansion_Group2 (CTCL Patients)
Number analyzed (Participants) | 2 | 2 | 0 | 7 | 6
days | 151 [65 to 151] | 151 [65 to 151] |  | 151 [65 to 151] | 114 [57 to 114]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Assessment of Cmax in subjects treated with Tenalisib and Romidepsin combination. Blood samples for measurement of RP6530 plasma concentrations were collected pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 10, and 11 hours after dosing on Day 8 of the first cycle. Maximum (peak) drug concentration (Cmax in nanograms/milliliter) was estimated using Single-Dose data.
Time Frame: 8 days
Population: Peak Plasma Concentration (Cmax) of RP6530 at Cycle 1 day 8.
Measure: Mean (Standard Deviation); unit: nanogram/millilitre
Arm/Group | Dose escalation_Cohort 1 | Dose escalation_Cohort 2 | Dose escalation_Cohort 3
Number analyzed (Participants) | 3 | 3 | 3
nanogram/millilitre | 1544.42 (1609.44) | 2152.17 (748.83) | 5791.11 (2426.44)

ADVERSE EVENTS:
Time Frame: 7 months
Description: Summary of Related Treatment-Emergent Adverse Events - All Patients. Patients were monitored for adverse events and both related and as well as non-related adverse events were captured during the study. The related adverse events (irrespective of single-agent or combination related) are reported here.
Arm/Group | Dose escalation_Cohort 1 | Dose escalation_Cohort 2 | Dose escalation_Cohort 3 | Dose expansion_Group 1 (PTCL) | Dose expansion_Group 2 (CTCL)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/12 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 1/12 | 2/12
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose escalation_Cohort 1 (N=3) | Dose escalation_Cohort 2 (N=3) | Dose escalation_Cohort 3 (N=3) | Dose expansion_Group 1 (PTCL) (N=12) | Dose expansion_Group 2 (CTCL) (N=12)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose escalation_Cohort 1 (N=3) | Dose escalation_Cohort 2 (N=3) | Dose escalation_Cohort 3 (N=3) | Dose expansion_Group 1 (PTCL) (N=12) | Dose expansion_Group 2 (CTCL) (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (5) | 2 (6) | 2 (7) | 8 (33) | 4 (11)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (5) | 0 (0) | 5 (24) | 2 (18)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (1) | 8 (10) | 12 (20)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Abdomial pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 3 (4) | 1 (1) | 1 (1) | 6 (6) | 7 (9)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 7 (21)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 6 (19)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (4)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 2 (7)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (4)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Blood Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (7)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03770000/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03770000/SAP_001.pdf